CLINICAL TRIAL: NCT06414447
Title: SANSA Electrocardiogram (ECG) Validation Study
Brief Title: Electrocardiogram (ECG) Validation Study
Status: Not yet recruiting | Type: Observational
Sponsor: Huxley Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-10000
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Arrythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Huxley Medical — diagnostic

SUMMARY:
Comparison of diagnostic Electrocardiogram (ECG) signals

ELIGIBILITY:
INCLUSION CRITERIA

* 18 years of age of older
* Able to read, understand, and sign informed consent documentation willing to wear the Sansa device and 3-lead or 5-lead Holter monitor simultaneously for 24- hours
* In the opinion of the investigator, subject is willing to comply with the protocol

EXCLUSION CRITERIA

* Noted deformities of the chest (e.g., pronounced scarring, pectus carinatum) that would Interfere with sensor placement
* broken or injured skin that would interfere with sensor placement, are known to experience adverse reactions to medical-grade adhesive
* pacemaker dependent
* females who are pregnant (self-reported)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects willing to participate in an ECG diagnostic evaluation
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of the diagnostic Electrocardiogram (ECG) signal quality of the P, QRS and T wave deflections of the Sansa device to a reference standard Holter monitor | 3 months